CLINICAL TRIAL: NCT04612062
Title: A First-in-Human Study to Determine Safety, Tolerability and Systemic Exposure of Topically Applied CEE321 Cream in Adult Subjects
Brief Title: A First-in-Human Study of CEE321 in Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCEE321A12101; jRCT2031200317 (Other: jRCT)
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Atopic Dermatitis
Keywords: First-in-Human; Healthy Volunteers; Atopic Dermatitis; CEE321; Safety; Tolerability; Pharmacokinetics
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: This is a FIH study of CEE321 in Adult Healthy Subjects (Part A) and Subjects with Atopic Dermatitis (Part B).
  Enrollment started with Healthy Subjects in Feb 2020. The protocol was amended Jul 2020 to include Atopic Dermatitis (AD) Subjects (Part B).
Masking Description: Open Label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Subjects (Part A) (Experimental): CEE321 0.2% (3 mg/cm2) topical cream b.i.d.
  Interventions: Drug: CEE321
- Atopic Dermatitis (Part B) (Experimental): CEE321 0.2% (3 mg/cm2) topical cream b.i.d.
  Interventions: Drug: CEE321

INTERVENTIONS:
Drug: CEE321 — CEE321 administered to all subjects
  Other Names: CEE321 0.2% (3 mg/cm2) topical cream b.i.d.

SUMMARY:
Open label, non-randomized, uncontrolled, First-in-Human Phase 1 Study in Healthy Subjects and Subjects with Atopic Dermatitis

ELIGIBILITY:
Key inclusion Criteria for Healthy Subjects (Part A)

* Written informed consent
* Able to communicate well with the investigator to understand and comply with the requirements of the study, including skin biopsies
* Healthy male and female subjects aged ≥18 and ≤ 65 years
* Able to comply with requirement of domiciliation at the investigational site

Key Exclusion Criteria for Healthy Subjects (Part A)

* Subjects with a history of hypertrophic scars or keloids.
* Any infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals and/or hospitalization, isolation, quarantine within 4 weeks prior to first treatment
* Women of childbearing potential defined as all women physiologically capable of becoming pregnant.
* History of drug or alcohol abuse within the 12 months prior to dosing

Key inclusion Criteria for Atopic Dermatitis Subjects (Part B)

* Written informed consent
* Able to communicate well with the investigator to understand and comply with the requirements of the study, including skin biopsies
* Adult male or female subjects aged ≥18 and ≤ 65 years with confirmed clinical diagnosis of atopic dermatitis (AD)

Key Exclusion Criteria Atopic Dermatitis Subjects (Part B)

* Subjects with a history of hypertrophic scars or keloids.
* Any infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals and/or hospitalization, isolation, quarantine within 4 weeks prior to first treatment
* Women of childbearing potential defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception
* History of drug or alcohol abuse within the 3 months prior to dosing
* Any skin disease that, in the opinion of the investigator, would confound the diagnosis or evaluation of AD disease activity
* Clinical significant medical condition, including psychiatric condition, which in the Investigator's opinion may interfere with safety of subjects, study objectives or adherence to the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | adverse events recorded during study

SECONDARY OUTCOMES:
Plasma trough concentration of CEE321 | day 15

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Novartis Investigative Site, Glendale, California
  - Novartis Investigative Site, Baltimore, Maryland
- Novartis Investigative Site, Hachiōji, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: jRCT — https://jrct.niph.go.jp/en-latest-detail/jRCT2031200317